CLINICAL TRIAL: NCT06772649
Title: Investigating the Safety and Efficacy of Compression Therapy for Controlling Swelling in Post-Injury Ankle Management
Brief Title: Compression Therapy for Swelling Management Following Ankle Injury
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Bauerfeind (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSWELL-001
Record Dates: First submitted 2025-01-09; First posted 2025-01-13 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Ankle Fracture; Ankle Arthrodesis
Keywords: non-operative ankle fracture management; operative ankle fracture management; ankle arthrodesis; mid-foot arthrodesis; hind-foot arthrodesis
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bauerfeind Ankle Compression Sleeve (Experimental): Patients in this arm will be fitted for a Bauerfeind ankle compression sleeve at 6 weeks post-injury/post-operative following the removal of their walking boot. Patients will use the compression sleeve until 6 months post-injury/post-operative.
  Interventions: Other: Compression sleeve
- Control (No Intervention): Patients in the control group will wear a walking boot until 6 weeks post-injury/post-operative. Upon removal of the boot, no swelling aid will be provided to patients (as per standard of care)

INTERVENTIONS:
Other: Compression sleeve — The Bauerfeind compression sleeve is a fabric sleeve designed to support the ankle during movement. It's made of a compressive knit material that increases sensorimotor feedback, enhances blood circulation, and stimulates metabolism. The design helps reduce ligament strain, activates the foot's stabilizing muscles more quickly, and improves joint coordination.
  Other Names: Bauerfeind ankle compression sleeve
  Arms: Bauerfeind Ankle Compression Sleeve

SUMMARY:
After an injury or undergoing foot/ankle surgery, patients often experience swelling in the injured area. Under current standard of care, plaster casts are removed at six weeks and patients are put in a walking boot. At this point in time of their recovery, patients are permitted to weight bear and move in their walking boot without other help, like crutches. This has shown to cause a significant amount of swelling in the ankle and foot between week six and twenty-six post-injury/surgery.

There is not much research that has looked at the effects of compression on reducing swelling in post-operative and non-operative ankle fracture, mid-foot, hindfoot, or ankle arthrodesis. This research is important because post-injury swelling can lead to wound complications and limit functionality. Therefore, finding new ways to reduce swelling could help prevent future complications.

The purpose of this study is to see if the Bauerfeind ankle compression sleeve is a safe post-operative/injury foot and ankle swelling management tool. Use of a compression sleeve will be compared to just using a walking boot, which is current standard of care, to determine if the compression sleeve reduces post-operative/injury foot and ankle swelling.

The study will follow patients improvement in swelling and pain. The compression sleeve will also be assessed for product safety. Safety is determined by watching the frequency, severity and seriousness of any side effects or complications, known as adverse events, that may be experienced while in the study.

The Bauerfeind ankle compression sleeve has been and is currently used in humans as a swelling reducing devise in the foot and ankle but has not been studied in a randomized control trial.

DETAILED DESCRIPTION:
This research study aims to assess swelling at 6, 12 and 26 weeks post non-operative and operative ankle fracture, mid-foot, hind-foot or ankle arthrodesis. Under current management, plaster casts are removed at six weeks and patients continue care in a walking boot. At this point in time of their recovery patients are permitted to weight bare and move in their walking boot without other aids. This has shown to cause a significant amount of swelling in the ankle and foot between week 6 and twenty-six post-injury/surgery.

To minimize swelling this study proposes the use of an ankle compression sleeve to wear during management once the plaster cast has been removed at 6 weeks. There is limited literature examining the effects of compression on reducing swelling in post-operative and non-operative ankle fracture, mid-foot, hindfoot, or ankle arthrodesis. This research is important as post ankle injury swelling can lead to wound complications and limit functionality. Thus, identifying management tools that reduce swelling may limit future complications.

Patients at the Queen Elizabeth II Health Sciences Centre that are undergoing non-operative ankle fracture management, ankle fracture surgery, or hind-foot, mid-foot, or ankle arthrodesis that meet the inclusion and exclusion criteria and willingly consent to the study will be included in the study's participant pool. Participants will be randomly assigned to control and intervention groups. Both groups will undergo a volume displacement swelling measurement of each foot at 6 weeks post operation/injury.

Patients in intervention group will be given a Bauerfeind ankle compression sleeve to wear under the walking boot for the rest of their management protocol. Patients will undergo volume displacement and compliance/ accessibility questionnaires during their twelve week and 6-month post operation/injury clinic visits. Data will be summarized and compared between groups and within groups at at 6, 12 and 26 weeks post operation/injury for change in swelling.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing outpatient ankle, mid-foot or hindfoot arthrodesis, fracture surgery, or non-operative ankle fracture management at the Queen Elizabeth II Health Sciences Center.
* Aged 18 or over

Exclusion Criteria:

* Patients undergoing other ankle procedures
* Patients who have any signs of wound healing complications post-surgery
* Patients who are unable to progress to walking boot and weight-bearing management at 6 weeks post operation/injury.
* Patients with other co-morbidities that may create bias within the results (lymphedema, heart conditions etc.)
* Patients who are unable to speak and read English, and/or in the opinion of the Principal Investigator are unable to provide fully informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Swelling (volume) | 6 weeks, 12 weeks, and 24 weeks post-injury/post-operative
  Ankle swelling will be measured using a standard volume displacement test. Patients will place their foot in a tub of water of known volume, and the displaced volume will be measured. This procedure will be completed for both ankles.

SECONDARY OUTCOMES:
Visual Analog Scale for Pain | 6 weeks, 12 weeks, and 24 weeks post-injury/post-operative
  Ankle pain will be measured using a standard Visual Analog Scale (VAS) to determine the level of pain a patient is experiencing.
Product-Related Safety | 6 weeks, 12 weeks, and 24 weeks post-injury/post-operative
  Safety of the Bauerfeind ankle compression sleeve will be determined by monitoring product-related adverse events. These could include things like skin irritation or reduced joint mobility due to use of the study product. All adverse events will be documented by severity and relationship to the study product.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth II Health Science Center, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No